CLINICAL TRIAL: NCT00896324
Title: Assessment and Treatment of Cognitive Deficits in Breast Cancer
Brief Title: Intellectual Impairment in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Oxana Palesh, Assistant Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IRB-14623 part 1; SU-04062009-2139 (Other: Stanford University); BRS0002 (Other: OnCore); NCT00866931 (obsolete NCT alias)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Cognitive Training; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Pre-chemotherapy participants are randomized between active neurofeedback, and a sham (placebo) neurofeedback.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Rehabilitation (Breast Cancer(BC) with chemotherapy) (Active Comparator): Cognitive rehabilitation is a very low-risk method of treatment for cognitive deficits that involves restoring impaired function and/or training the individual to compensate for the area of deficit. Subjects will complete a curriculum of cognitive exercises 30 minutes per day, 5 days per week for 6-weeks.
  Interventions: Behavioral: Cognitive Rehabilitation
- Active Neurofeedback (BC pre-chemotherapy) (Active Comparator): In active Neurofeedback session subjects will be trained to increase brain activation in regions associated with executive function (EF) function deficits (as determined by neuroimaging measures) by viewing their own brain activation in real-time. The "dose" will be 2-3 sessions, each lasting approximately 30 minutes.
  Interventions: Behavioral: Active Neurofeedback Training
- Neurofeedback placebo (Sham) (BC pre-chemotherapy) (Sham Comparator): Neurofeedback training: 2-3, 30 min training sessions. For the sham placebo group, fabricated real-time data will be provided to the subject as feedback information hence enabling the subject to view information identical to experimental subjects but without accurate data pertaining to their own brain activation. The technician will be blinded to the subject's treatment condition assignment.
  Interventions: Behavioral: Neurofeedback Training (placebo / Sham)

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — The cognitive rehabilitation procedure will involve a curriculum of game-like cognitive exercises designed to facilitate graded practice of EF skills including attention, processing speed, mental flexibility, planning and logic. The exercises will be delivered to participants via a secure, password protected website created specifically for this study by the PI. Subjects will complete a curriculum of cognitive exercises 30 minutes per day, 5 days per week for 6-weeks.
  Arms: Cognitive Rehabilitation (Breast Cancer(BC) with chemotherapy)
Behavioral: Active Neurofeedback Training — Neurofeedback training is a type of biofeedback during which the subjects will be trained to improve cognitive function by implementing certain cognitive strategies while receiving feedback of their own brain activity. This is done using an infrared spectroscopy (NIRS) system. NIRS measurements will be performed using an ETG-4000 NIRS system (Hitachi Medical, Tokyo, Japan), at two wavelengths of near-infrared light (695 and 830 nm). Each participant will have 2 or 3 sessions, each lasting approximately 30 minutes.
  Arms: Active Neurofeedback (BC pre-chemotherapy)
Behavioral: Neurofeedback Training (placebo / Sham) — Neurofeedback training: 2-3, 30 min training sessions. For the sham placebo group, fabricated real-time data will be provided to the subject as feedback information hence enabling the subject to view information identical to experimental subjects but without accurate data pertaining to their own brain activation. The technician will be blinded to the subject's treatment condition assignment.
  Arms: Neurofeedback placebo (Sham) (BC pre-chemotherapy)

SUMMARY:
RATIONALE: Breast cancer and its treatment may cause changes in a patient's ability to think, learn, and remember. Gathering information about a woman's genes, brain function, and personal history may help doctors learn more about the disease and plan the best treatment.

PURPOSE:

1. To determine changes in brain function that occur following breast cancer chemotherapy.
2. To gain further understanding of the individual differences in brain function changes and recovery based on demographic, medical and treatment variables.

DETAILED DESCRIPTION:
This study aims to determine some of the genetic, neurobiologic and demographic factors that are associated with cognitive outcome following breast cancer (BC). Additionally, it aims to test novel behavioral interventions designed to improve executive function skills following BC treatment.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Primary, non-metastatic breast cancer

3.1.2 Newly diagnosed patients who have not yet begun treatment.

3.1.4 Female participants age 40-65 years of all ethnicities who speak fluent English will be recruited.

3.1.5 There are no life expectancy restrictions.

3.1.6 Karnofsky Performance Status 70% minimum. ECOG will not be employed.

3.1.7 There are no requirements for marrow function. The brain must be free from gross neuropathology and metastases in order to participate.

3.1.8 Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2.1 History of cognitive, psychiatric or medical conditions prior or unrelated to cancer diagnosis and/or known to significantly impact assessments (e.g. premature birth, developmental delays, learning disabilities, severe psychiatric conditions, brain injury, stroke). Non-English speaking. Major sensory impairment (e.g. hearing loss, blindness) that would render assessments invalid. MRI contraindications (e.g. metallic implants or devices). Distant metastases. See also section 4.2.1.

3.2.2 Participants currently involved in studies specifically aimed at improving cognitive symptoms will be excluded.

3.2.3 Participants with significant co-morbid diseases known to significant impact neuropsychological function such as Alzheimer's or Parkinson's will be excluded.

3.2.4 There are no known risks for allergic reactions to any of the study procedures.

3.2.5 Participants taking certain medications that affect neuropsychological and/or brain function including Haldol, Aricept, Ritalin, etc. will be excluded. Most anti-depressants are acceptable. Some anti-anxiety medications may not be. Each case will be individually reviewed.

3.2.6 There are no other agent-specific exclusion criteria.

3.2.7 Pregnant individuals will be excluded as this is a contraindication for the 3 Tesla research MRI scanner employed by this study but not because of the treatment programs per se. Nursing individuals can enroll.

3.2.8 Patients who are HIV positive will be excluded given the known effects of this condition on cognitive function which would confound the effects of anti-cancer treatments on cognitive outcome.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01-12 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Examine the effectiveness of a cognitive rehabilitation program for improving executive function (EF) deficits for preventing or lessening EF impairments in women with Breast Cancer | 6 weeks
  Evaluation of efficacy of executive function (EF) will be done via Neuropsychological and Neuroimaging (using functional MRI) assessments. Measurements of executive function, memory, processing speed, attention, visual-spatial processing and language will be compared before and after 6 weeks of cognitive rehabilitation program. Neuropsychological assessment and neuroimaging assessment changes will be compared from baseline to post-assessment in the intervention groups. Mixed effects approach and reliable change index (RCI) will be used as a supplementary analysis to determine the change in cognitive testing scores from pre- to post-intervention.Specific neuroimaging data (e.g. prefrontal cortex volumes, hippocampal metabolite levels, whole brain white matter fractional anisotropy) will be correlated with neuropsychological testing scores.

SECONDARY OUTCOMES:
Examine the effectiveness of neurofeedback training program for preventing or reducing cognitive deficits in women with Breast Cancer | up to 6 months
  Neurofeedback training test will be done on women with BC, prior to receiving adjuvant chemotherapy. For the sham placebo group, fabricated real-time data will be provided to the subject as feedback information. Prefrontal and parietal regions of interest will be measured by putting a nylon cap attached to 16 optode emitter/receiver pairs on each subject's head covering the bilateral frontal and parietal regions symmetrically. Measurements will be recorded every 0.1s. The pretask baseline will be determined
Evaluate diurnal cortisol levels on executive function outcome in women with Breast cancer | 2 days
  Saliva collection for cortisol analysis will be done with women with BC/chemotherapy, women BC/ no chemotherapy and healthy women. Saliva samples for cortisol analysis will be collected from subjects on 2 consecutive days after the neuropsychological testing and MRI scan have been completed using SARSTEDT Salivettes. Cortisol analysis will be conducted using luminescence immunoassay. The cortisol slope of baseline days will be used as a measure of baseline cortisol level. Cortisol Levels will be correlated with cognitive testing scores.

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Palesh, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No